CLINICAL TRIAL: NCT05127694
Title: Comparison of the Efficacy of Medical Treatment and Vestibular Rehabilitation In Patients With Acute Benign Paroxysmal Positional Vertigo
Brief Title: Treatment In Acute Benign Paroxysmal Positional Vertigo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, gorkem ata, Physiotherapist MSc, Lecturer, Medipol University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10840098-604.01.01-E.19383
Record Dates: First submitted 2021-10-06; First posted 2021-11-19 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Benign Paroxysmal Positional Vertigo; Balance; Distorted; Vestibular Disorder; Dizziness
Keywords: Benign Paroxsymal Positional Vertigo; Balance; Pysiotherapy and Rehabilitation; Canalith Repositioning Procedure; Pharmacological Therapy; Dynamic Visual Acuity; Dizziness
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo; Vestibular Diseases; Dizziness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vestibular Rehabilitation Group (Experimental): Investigators applied vestibular rehabilitation in this group. This group was consist of 15 participants. After the evaluation investigators gave the patients repetitive vestibular exercises for 4 weeks and in the first week investigators performed canalith repositioning procedure depending on the affected canal. If affected posterior semicircular canal investigators applied Epley maneuver. If affected horizontal semicircular canal also applied barbeque roll maneuver.
  Interventions: Other: Vestibular Rehabilitation
- Pharmacological Control Group (No Intervention): Investigators did not apply any treatment in this group. Participant in this group just used medications doctor-prescribed.

INTERVENTIONS:
Other: Vestibular Rehabilitation — Vestibular Rehabilitation which is consist of repetitive exercises and canalit repositioning maneuvers
  Arms: Vestibular Rehabilitation Group

SUMMARY:
Benign paroxysmal positional vertigo (BPPV) is a vestibular disorder that manifests itself as a result of dizziness caused by the otoconia in the inner ear coming out of their places and circulating freely in the semicircular canals or by attaching to the cupula and sensitizing the cupula to head movements against gravity. The aim of the study is to compare the effectiveness of pharmacological treatment initiated by the physician and vestibular rehabilitation initiated by physiotherapist in patients with acute benign paroxysmal positional vertigo (BPPV). Thirty patients, aged 18-50 years, who applied to the Bağcılar Safa Hospital, were included in the study. The patients were divided into two groups, 15 pharmacological control group and 15 vestibular rehabilitation group. 8 patients in the pharmacological control group were given the drug containing betahistine by the physician, and 7 patients received the drug containing additional dimenhydrinate to the betahistine. In the rehabilitation group, exercises including head and eye movements and maneuvering were performed according to the direction of the canal after the exercise, and the patients were given a home exercise program. Treatment continued for 4 weeks. Visual Analogue Scale (VAS), dynamic visual acuity test, romberg, semitandem, tandem posture tests with a stopwatch, standing test on one leg with eyes open and closed, and unterberger tests were applied to patients before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years of age,
* Positive Dix-Hallpike test result, and
* No spontaneous nystagmus.

Exclusion Criteria:

* Patients with Meniere's disease, vestibular neuritis, labyrinthitis, sudden sensory hearing loss, chronic otitis media, non-ambulatory patients, patients with vertigo due to central causes, and patients with cardiac complaints were excluded from the study.
* In addition, patients with conditions contraindicated for canalith repositioning procedures (such as cervical spine stenosis, severe kyphoscoliosis, cervical radiculopathy, ankylosing spondylitis, severe lumbar dysfunction, and spinal injuries) were excluded from the vestibular rehabilitation group.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-12-08 (Actual); Study Completion 2020-04-16 (Actual)

PRIMARY OUTCOMES:
Perceptual Dizziness | Four weeks
  Perceived dizziness was assessed using the Visual Analog Scale (VAS). The patients stated the severity of their dizziness between 0-10 (0 being the mildest, 10 being unbearable).
Balance | Four weeks
  The balance of the patients was evaluated using the tandem, romberg, and one-leg standing test with eyes open and closed using a stopwatch. Individuals were expected to maintain their balance for 30 seconds.
Vestibular Dysfunction | Four weeks
  Vestibular Dysfunction was assessed with the Unterberger Test performed with the eyes closed. During the Unterberger test, the patient should marching where they are. If more than 45 degrees of deflection is detected, the test is positive.
Dynamic Visual Acuity | Four weeks
  Dynamic visual acuity was evaluated using the Snellen chart. A person taking the test is seated in a chair 2 meters away from the Snellen chart and while the therapist shakes the patient's head from right to left, the patient is asked if he can see the letters of each line, starting from the top. The test is terminated on the line where the letter sequence cannot be seen clearly.

CONTACTS AND LOCATIONS:
Locations (1):
- Safa Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No